CLINICAL TRIAL: NCT04721639
Title: Effect of Sphinx Pose (Salamba Bhujangasana) Among Health Care Providers With Chronic Low Back Pain: A Randomized Controlled Trial.
Brief Title: To Observe the Effect of Sphinx Pose (Salamba Bhujangasana) Among Health Care Providers With Chronic Low Back Pain
Acronym: CLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Responsible Party: Principal Investigator, Shamoon Noushad, Principal Investigator, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PPL-SPHINX2020
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic Low back pain; Yoga therapy; Sphinx Pose Yoga (Salamba Bhujangasana).; Healthcare Providers; Substance P; Cortisol; Beta Endorphins

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental intervention (Sphinx Yoga Therapy) (Experimental): In this group, participants will be intervened with Sphinx Yoga therapy which will take place in a conserved therapy center of Koohi Goth Hospital. This stretching exercise session will take place in the afternoon and for a duration of 10 minutes followed by 30 minutes therapy session five times per week (total 12 weeks).
  Interventions: Other: Sphinx Yoga Therapy
- The control intervention (Usual Care) (No Intervention): In this Group, participants won't be receiving any intervention and provided with the usual care.

INTERVENTIONS:
Other: Sphinx Yoga Therapy — Sphinx Pose Yoga is among the best beginner Yoga Poses that relieve Lower Back Pain. It extends the back gently and activates muscles along the spine. The subject will be asked to lay down on their stomach with feet set hip-width apart, the elbows positioned under the shoulders, and the legs held together. The chin should be pointing towards the floor. Next, the subject is required to pull up the kneecaps, squeezing the thighs and buttocks, pressing the pubic bone into the floor and dropping shoulders back away from the neck and pushing the chest forward. In this position, the subject is asked to breathe and hold the pose for two to six breaths. By the end, the subject will be required to exhale, bringing the elbows to the sides and slowly lowering the chest and head to the floor.
  Arms: The experimental intervention (Sphinx Yoga Therapy)

SUMMARY:
This Randomized Controlled trial is designed to observe the effect of Sphinx Yoga (Salamba Bhujangasana) on low back pain and variation in the associated physiological parameters that help explain the beneficial effects of yoga, among healthcare providers of Karachi Pakistan. Healthcare providers with LBP (determined as per the baseline assessment) will be recruited and Substance P and Beta Endorphins will be assessed at baseline and after 3 months. The subjects with LBP will be determined based on the scores of the Oswestry Low Back Pain Disability Questionnaire, Numerical Pain Rating (NPR) scale, Roland Morris Disability Questionnaire (RMDQ) and Fear Avoidance Beliefs Questionnaire (FABQ) work subscale. Subjects meeting eligibility criteria will be randomly allotted to intervention and control groups. The study outcomes will be monitored in subjects of both groups at baseline and after 3-month follow-up (post-interventional).

DETAILED DESCRIPTION:
Plan of work

* Assessment of eligibility & Enrollment: HCPs experiencing LBP as per the eligibility criteria will be enrolled.
* Baseline Assessment: All the variables, i.e. Oswestry Low Back Pain Disability Questionnaire, World Health Organization Quality of Life (WHOQOL), Roland Morris Disability Questionnaire (RMDQ) and Sadaf Stress Scale (SSS), Substance-P and Beta Endorphins will be measured at baseline.
* Randomization & Allocation: Eligible consenting subjects will be randomly allocated to the experimental or control group.
* Follow-up Assessment: All the outcome measures observed at baseline will be re-assessed after 3 months.
* Statistical Analysis: Pre & post-analysis will be conducted.

Study design The study will be conducted as a Randomized Controlled trial at a primary healthcare setting. The participant eligibility will be assessed using a pre-screening questionnaire including components of disability questionnaires. Based on the eligibility criteria, consenting HCPs will be recruited and randomized into two groups i.e. Group A (experimental) including participants who will receive the intervention and Group B (control) receiving no intervention. The study outcomes will be monitored among participants of both groups at baseline and post-intervention (3-month follow-up).

Participants Healthcare providers with LBP will be recruited with no restriction for ethnicity or race. The participants from diverse socio-cultural backgrounds will be considered eligible if they meet the inclusion criteria. The study objective will be explained and participants will be invited to participate based on their free-will.

Sampling Size The required sample size for the two study groups with α = 0.05 and (1- α) = 0.80, was estimated to be 49 in each group i.e. the total sample size was 98 for two groups. The sample size calculator provided by the UCSF CTSI was used.

Randomization After assessing the eligibility the participants will be randomly allocated in the ratio of 1:1 to the study groups (experimental and control). The randomization sequence will be computer-generated. After acquiring the basic information, a unique code will be assigned to each of the study participants which will then be mentioned in their Performa.

Interventions • The experimental intervention: The Group A participants will be intervened with Sphinx Yoga therapy which will take place in a conserved therapy center of Koohi Goth Hospital. This stretching exercise session will take place in the afternoon and for a duration of 10 minutes followed by 30 minutes therapy session five times per week (total 12 weeks).

• The control intervention: Group B participants won't be receiving any intervention and provided with the usual care.

ELIGIBILITY:
Inclusion Criteria: All subjects must meet all the requirements as follow:

* Subjects of both genders between 25 to 45 years of age.
* They must score more than or equal to 2 for their pain intensity in the last week, on the Numerical Pain Rating (NPR) scale (0-10)
* On Roland Morris Disability Questionnaire participant's score should be ≥ 4.
* Fear Avoidance Beliefs Questionnaire (FABQ) work subscale score must be less than 19.
* They have visited the health care provider in recent days for their back pain.

Exclusion Criteria:

* Subjects with a personal history of neurological disorders including Alzheimer's, amyotrophic lateral sclerosis, multiple sclerosis, Parkinson's and stroke, any cardio-respiratory disorders like congestive heart failure, heart attack in the past 24 months and/or musculoskeletal disorders like rheumatoid arthritis, pathologic fractures of the spine, avascular necrosis or osteonecrosis, severe osteoarthritis. Including a history of spine surgery or hip arthroplasty.
* Those subjects who have used narcotics or muscle relaxants within 30 days prior to study enrollment.
* Pregnant and/or lactating females.
* Those having body mass index > 35 kg/m2 or presented with unexplained weight loss over the past month (>10 lbs).
* Clinically depressed subjects (i.e., subjects who score 24 or higher on the Center for Epidemiology Depression Scale).

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Extent of Disability | 3 Months
  Change in the Oswestry Disability Index will be observed among the subjects enrolled in the experimental group after intervention. The Oswestry Low Back Pain Disability Questionnaire, is considered as a standard to assess the functionality of low back. It is considered a gold standard tool for evaluating the extent of disability.
Pain Score | 3 Months
  It will be assessed with the help of Numeric Pain Rating scale. The numeric rating scale is a pain screening tool that is frequently used to evaluate the current level of pain using a 0-10 scale, where 0 corresponds to "no pain" and 10 to "the greatest pain possible."

SECONDARY OUTCOMES:
Substance P | 3 Months
  Change in the Substance P level will be observed among the subjects enrolled in the experimental group as compared to the control group
Beta Endorphins | 3 Months
  Change in the Beta Endorphins level will be observed among the subjects enrolled in the experimental group as compared to the control group
Cortisol | 3 Months
  Change in the Cortisol level will be observed among the subjects enrolled in the experimental group as compared to the control group
Quality of Life Score | 3 Months
  Change in World Health Organization Quality of Life (WHOQOL) from baseline to post-intervention assessment. It will help in the evaluation in changes observed in the well-being of the patient, before and after the intervention is given.
Physical Stress - Stress Score | 3 Months
  SSS was established for stress evaluation by observing major signs & symptoms, and classification of these symptoms into seven different classes47. Physical stress, sub-section of SSS will be used to assess the degree of stress and its contribution in LBP.

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Koohi Goth Women Hospital, Karachi, Sindh
  - Koohi Goth Women Hospital, Karachi, Sindhi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patil NJ, Nagaratna R, Tekur P, Manohar PV, Bhargav H, Patil D. A Randomized Trial Comparing Effect of Yoga and Exercises on Quality of Life in among nursing population with Chronic Low Back Pain. Int J Yoga. 2018 Sep-Dec;11(3):208-214. doi: 10.4103/ijoy.IJOY_2_18. PMID 30233114
- [Background] Sherman KJ, Cherkin DC, Cook AJ, Hawkes RJ, Deyo RA, Wellman R, Khalsa PS. Comparison of yoga versus stretching for chronic low back pain: protocol for the Yoga Exercise Self-care (YES) trial. Trials. 2010 Mar 31;11:36. doi: 10.1186/1745-6215-11-36. PMID 20356395
- [Background] Wieland LS, Skoetz N, Pilkington K, Vempati R, D'Adamo CR, Berman BM. Yoga treatment for chronic non-specific low back pain. Cochrane Database Syst Rev. 2017 Jan 12;1(1):CD010671. doi: 10.1002/14651858.CD010671.pub2. PMID 28076926
- [Background] Saper RB, Lemaster C, Delitto A, Sherman KJ, Herman PM, Sadikova E, Stevans J, Keosaian JE, Cerrada CJ, Femia AL, Roseen EJ, Gardiner P, Gergen Barnett K, Faulkner C, Weinberg J. Yoga, Physical Therapy, or Education for Chronic Low Back Pain: A Randomized Noninferiority Trial. Ann Intern Med. 2017 Jul 18;167(2):85-94. doi: 10.7326/M16-2579. Epub 2017 Jun 20. PMID 28631003
- [Background] Chang DG, Holt JA, Sklar M, Groessl EJ. Yoga as a treatment for chronic low back pain: A systematic review of the literature. J Orthop Rheumatol. 2016 Jan 1;3(1):1-8. PMID 27231715
- [Background] Behisi MA, Al-Otaibi ST, Beach J. Back pain among health care workers in a Saudi Aramco facility: prevalence and associated factors. Arch Environ Occup Health. 2013;68(1):30-8. doi: 10.1080/19338244.2011.627895. PMID 23298422
- [Background] Galantino ML, Bzdewka TM, Eissler-Russo JL, Holbrook ML, Mogck EP, Geigle P, Farrar JT. The impact of modified Hatha yoga on chronic low back pain: a pilot study. Altern Ther Health Med. 2004 Mar-Apr;10(2):56-9. PMID 15055095
- [Background] Simsek S, Yagci N, Senol H. Prevalence of and risk factors for low back pain among healthcare workers in Denizli. Agri. 2017 Apr;29(2):71-78. doi: 10.5505/agri.2017.32549. PMID 28895982
- [Background] Menzel N, Feng D, Doolen J. Low Back Pain in Student Nurses: Literature Review and Prospective Cohort Study. Int J Nurs Educ Scholarsh. 2016 May 13;13:/j/ijnes.2016.13.issue-1/ijnes-2015-0057/ijnes-2015-0057.xml. doi: 10.1515/ijnes-2015-0057. PMID 27176750
- [Background] Cinar-Medeni O, Elbasan B, Duzgun I. Low back pain prevalence in healthcare professionals and identification of factors affecting low back pain. J Back Musculoskelet Rehabil. 2017;30(3):451-459. doi: 10.3233/BMR-160571. PMID 27858698
- [Background] Mekonnen TH, Yenealem DG. Factors affecting healthcare utilization for low back pain among nurses in Gondar town, northwest Ethiopia, 2018: a cross-sectional study. BMC Res Notes. 2019 Mar 29;12(1):185. doi: 10.1186/s13104-019-4231-2. PMID 30922383
- [Background] Choi HY, Lee CH. Can Beta-Endorphin Be Used as a Biomarker for Chronic Low Back Pain? A Meta-analysis of Randomized Controlled Trials. Pain Med. 2019 Jan 1;20(1):28-36. doi: 10.1093/pm/pny186. PMID 30256990
- [Background] Parris WC, Kambam JR, Naukam RJ, Rama Sastry BV. Immunoreactive substance P is decreased in saliva of patients with chronic back pain syndromes. Anesth Analg. 1990 Jan;70(1):63-7. doi: 10.1213/00000539-199001000-00010. PMID 1688690
- [Background] Jasim H, Carlsson A, Hedenberg-Magnusson B, Ghafouri B, Ernberg M. Saliva as a medium to detect and measure biomarkers related to pain. Sci Rep. 2018 Feb 19;8(1):3220. doi: 10.1038/s41598-018-21131-4. PMID 29459715
- [Background] Murtezani A, Hundozi H, Orovcanec N, Sllamniku S, Osmani T. A comparison of high intensity aerobic exercise and passive modalities for the treatment of workers with chronic low back pain: a randomized, controlled trial. Eur J Phys Rehabil Med. 2011 Sep;47(3):359-66. Epub 2011 May 23. PMID 21602759
- [Background] Lisowska B, Lisowski A, Siewruk K. Substance P and Chronic Pain in Patients with Chronic Inflammation of Connective Tissue. PLoS One. 2015 Oct 7;10(10):e0139206. doi: 10.1371/journal.pone.0139206. eCollection 2015. PMID 26444559
- [Background] Kallman TF, Ghafouri B, Backryd E. Salivary beta-endorphin and substance P are not biomarkers of neuropathic chronic pain propensity. Heliyon. 2018 Aug 3;4(8):e00718. doi: 10.1016/j.heliyon.2018.e00718. eCollection 2018 Aug. PMID 30116793
- [Background] Zieglgansberger W. Substance P and pain chronicity. Cell Tissue Res. 2019 Jan;375(1):227-241. doi: 10.1007/s00441-018-2922-y. Epub 2018 Oct 3. PMID 30284083
- [Background] Noushad S, Ansari B, Ahmed S. Effect of nature-based physical activity on post-traumatic growth among healthcare providers with post-traumatic stress. Stress Health. 2022 Oct;38(4):813-826. doi: 10.1002/smi.3135. Epub 2022 Feb 26. PMID 35191173
- [Background] Noushad S, Ahmed S, Ansari B, Mustafa UH, Saleem Y, Hazrat H. Physiological biomarkers of chronic stress: A systematic review. Int J Health Sci (Qassim). 2021 Sep-Oct;15(5):46-59. PMID 34548863